CLINICAL TRIAL: NCT03180268
Title: Phase III Trial of Observation Versus Irradiation for a Gross Totally Resected Grade II Meningioma
Brief Title: Observation or Radiation Therapy in Treating Patients With Newly Diagnosed Grade II Meningioma That Has Been Completely Removed by Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN003; NCI-2016-01619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN003; NRG-BN003 (Other: NRG Oncology); NRG-BN003 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Grade 2 Meningioma; Intracranial Meningioma
MeSH Terms: conditions — Meningioma | interventions — Specimen Handling; Watchful Waiting; Observation; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (observation) (Active Comparator): Patients undergo observation. Additionally, patients undergo MRI and blood collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Clinical Observation; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment
- Arm II (radiation therapy) (Experimental): Patients undergo IMRT or proton beam radiation therapy 5 days a week over 6.5-7 weeks for a total of 33 fractions in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI and blood collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Clinical Observation — Undergo observation
  Other Names: observation
  Arms: Arm I (observation)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm II (radiation therapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
  Other Names: External beam radiation therapy protons (procedure); External Beam Radiotherapy (protons); PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; PROTON Therapy; Radiation, Proton Beam
  Arms: Arm II (radiation therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies how well radiation therapy works compared with observation in treating patients with newly diagnosed grade II meningioma that has been completely removed by surgery. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the extent of clinical benefit of the addition of adjuvant radiotherapy (RT) to gross total resection (GTR) for patients with newly diagnosed World Health Organization (WHO) grade II meningioma.

SECONDARY OBJECTIVES:

I. Overall survival (OS). II. Disease-specific survival (DSS). III. Toxicity (grade 3+, exclusive of expected alopecia). IV. Neurocognitive function (NCF). V. Patient reported outcomes (PRO) measurements. VI. Adherence to protocol-specific target and normal tissue parameters. VII. Concordance measurements of central versus parent-institution pathology. VIII. Assessment of pHH3 mitotic index and its correlation with progression-free survival (PFS) and OS.

IX. Validation of the prognostic value of a 34-gene expression biomarker. X. Validation of the predictive value of a 34-gene expression biomarker in predicting the benefit of radiotherapy.

XI. Tissue and specimen collection for future translational research.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo observation. Additionally, patients undergo magnetic resonance imaging (MRI) and blood collection throughout the study.

ARM II: Patients undergo intensity-modulated radiation therapy (IMRT) or proton beam radiation therapy 5 days a week over 6.5-7 weeks for a total of 33 fractions in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI and blood collection throughout the study.

After completion of study treatment, patients are followed up at 3, 6, and 12 months, every 6 months for year 2 and 3, then yearly for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* The patient must have a newly diagnosed unifocal intracranial meningioma, gross totally resected, and histologically confirmed as WHO grade II based upon pathology findings at the enrolling institution. WHO grade will be assigned according to WHO 2016 criteria
* Gross total resection (GTR) will be interpreted as modified Simpson grade 1-3 without gross residual dural-based or extradural tumor. GTR must be confirmed both by modified Simpson grade and by post-operative magnetic resonance imaging (MRI) findings. The modified Simpson grade can be inferred from the operative report (surgeon does not need to explicitly describe the Simpson grade for the purposes of eligibility)
* Step 1 registration must occur within 180 days of the initial surgery; this will provide sufficient time for post-operative imaging confirmation of resection extent after resolution of operative changes. Moreover, it will permit additional surgery if needed to achieve a GTR. Within this 180 day interval, a second surgery is permitted in order to achieve GTR, but even with a second surgery, Step 1 registration must occur within 180 days of the initial resection
* GTR must be confirmed on post-operative imaging following the most recent surgery. For protocol enrollment, the assessment of GTR will be made at each site. However, submission of both pre-operative and post-operative MRIs is required for patients. If a second surgery is performed, submission of post-operative MRI is required and pre-operative MRI is required only if obtained. All sequences obtained in the pre- and post-operative MR imaging are to be submitted to National Radiology Group (NRG) Oncology for study registration. The post-operative MRI must be completed within sufficient time to permit step 1 registration within 180 days of the initial resection. These same conditions apply in the setting of a second surgical procedure, although if a second surgery is completed, step 1 registration must still occur with 180 days of initial surgery. Computed tomography (CT) imaging is not required, but may be obtained if desired clinically, for instance to assess calcifications or hyperostosis
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* NOTE: Central pathology review must occur between steps 1 and 2 of registration. Once appropriate pathology specimens are received, central pathology review will occur within 10 business days, and must confirm WHO grade II meningioma before the patient can proceed to step 2 registration and randomization
* PRIOR TO STEP 2 REGISTRATION:
* Histologically confirmed diagnosis of WHO grade II meningioma confirmed by central pathology review prior to step 2 registration
* Age >= 18
* History/physical examination, including neurologic examination within 60 days prior to step 2 registration
* Post-operative Zubrod performance status 0-1 within 60 days prior to step 2 registration
* If the patient is a woman is of childbearing potential, a serum pregnancy test, obtained within 14 days prior to step 2 registration, must be negative, and, if randomized to receive radiation therapy, the woman must agree to use contraception

Exclusion Criteria:

* Optic nerve sheath meningioma, spinal or other extracranial meningioma, multiple meningiomas, hemangiopericytoma
* Definitive evidence of metastatic meningioma (metastasis, although rare, can occur and is exclusionary)
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (carcinoma in situ of the breast, oral cavity, cervix, melanoma in situ, or other non-invasive malignancies are permissible)
* Previous radiotherapy to the scalp, cranium, brain, or skull base and radiation-induced meningiomas
* Major medical illnesses or psychiatric impairments, which in the investigators opinion, will prevent administration or completion of the protocol therapy and/or preclude informed consent; these include, but are not restricted to:

  * Unstable angina and/or congestive heart failure requiring hospitalization at the time of step 2 registration
  * Transmural myocardial infarction within the last 6 months prior to step 2 registration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of step 2 registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of step 2 registration
  * Type II neurofibromatosis (NF2)
  * Ailments entailing substantial increases in sensitivity and side effect risk from radiation therapy (ataxia telangiectasia, Nijmegen breakage syndrome, and human immunodeficiency virus (HIV) with CD4 count < 200 cells/microliter); HIV testing is not required for eligibility for this protocol, and known HIV positive patients are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to step 2 registration
  * Inability to undergo MRI with and without contrast (e.g. claustrophobia, non-MRI compatible implant or foreign body, gadolinium allergy or renal dysfunction preventing the patient from receiving gadolinium- institutional guidelines should be used to determine if patients are at risk for renal dysfunction). Note that patients with severe claustrophobia are permitted on this study if they are willing and able to undergo MRI with adequate sedation or anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization to the first documented disease progression, or death due to any cause, whichever comes first, assessed up to 10 years
  Kaplan-Meier method will be used to calculate the PFS rates for each of the two arms. Hazard ratio (HR) on the treatment effect will be calculated using the Cox proportional hazard model. A one-sided log-rank test will be used to test the difference in PFS between the two arms.

SECONDARY OUTCOMES:
PFS | From randomization to the first documented disease progression, or death due to any cause, whichever comes first, assessed at 3 years
  Will be calculated based on the Kaplan-Meier curve. Cox proportional hazard model will be used to determine the adjusted treatment effect on PFS, with patient pretreatment characteristics as covariates.
PFS | From randomization to the first documented disease progression, or death due to any cause, whichever comes first, assessed up to 5 years
  Will be calculated based on the Kaplan-Meier curve. Cox proportional hazard model will be used to determine the adjusted treatment effect on PFS, with patient pretreatment characteristics as covariates.
Disease-specific survival (DSS) | From randomization to disease-related death, assessed up to 10 years
  Will be calculated using the cumulative incidence function for each arm. The HR for the treatment effect on DSS will be calculated using Gray's method under the competing risk approach, with death due to non-disease related cause treated as the competing risk. Multivariate analysis on DSS will be performed using the Fine-Gray model, with patient pretreatment characteristics as covariates.
DSS rates | At 3 years
  Will be calculated using the cumulative incidence function for each arm. The HR for the treatment effect on DSS will be calculated using Gray's method under the competing risk approach, with death due to non-disease related cause treated as the competing risk. Multivariate analysis on DSS will be performed using the Fine-Gray model, with patient pretreatment characteristics as covariates.
DSS rates | At 5 years
  Will be calculated using the cumulative incidence function for each arm. The HR for the treatment effect on DSS will be calculated using Gray's method under the competing risk approach, with death due to non-disease related cause treated as the competing risk. Multivariate analysis on DSS will be performed using the Fine-Gray model, with patient pretreatment characteristics as covariates.
Overall survival (OS) | From randomization to death due to any cause, assessed up to 10 years
  Cox proportional hazard model will be used to determine the adjusted treatment effect on OS, with patient pretreatment characteristics as covariates.
OS rates | At 5 years
  Will be calculated based on the Kaplan-Meier curve. Cox proportional hazard model will be used to determine the adjusted treatment effect on OS, with patient pretreatment characteristics as covariates.
Incidence of adverse events (exclusive of alopecia) | Up to 3 years
  Will be measured by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4 (version 5 beginning April 5, 2018).
Adherence rate to protocol-specific target and normal tissue parameters | Up to 10 years
Concordance rate of central versus parent-institution pathology | Up to 10 years
Prognostic value of 34-gene expression biomarker | Up to 5 years
  Will generate Kaplan-Meier curves for different risk subgroups defined by the risk scores, separately for post-operative observation and post-operative radiotherapy arms. The log-rank test will be used to test the difference in clinical outcomes (PFS and OS) between molecular risk subgroups (separately for the post-operative observation arm and post-operative radiotherapy arm). Cox proportional hazard model will be used to estimate the prognostic effect of the gene expression defined risk groups on clinical outcomes adjusting for pre-treatment patient characteristics as well as treatment arm.
Predictive value of 34-gene expression biomarker | Up to 5 years
  Will be evaluated formally through the test of a statistical interaction between molecular risk group (low/intermediate versus high) and treatment (observation versus radiotherapy). The Kaplan-Meier curves of PFS and OS between treatment arms will be displayed separately among low/intermediate risk and high-risk groups. A Cox proportional hazards model will be built including treatment group, gene expression risk group, an interaction term between treatment and gene expression risk group, as well as other pre-treatment patient characteristics. The interaction test will be based on a two-sided 0.05 level Wald test in the Cox proportional hazards model. The treatment difference between radiation therapy and observation will also be tested within each gene expression risk subgroup in a multivariable Cox proportional hazards model, adjusting for other patient characteristics.
Change in neurocognitive function (NCF) assessed by MD Anderson Symptom Inventory with Brain Tumor (MDASI-BT) | Baseline up to 60 months
  Will use a 2-sample t-test with a one-sided significance level of 0.05, with a Bonferroni adjustment to account for the neurocognitive function and symptom assessments resulting in an overall type I error of 0.1, there will be 72% statistical power to detect a medium effect size of 0.5 standard deviation (SD) for a comparison of the change from baseline to 6 months after randomization between the experimental and the control arm. Will compare NCF outcomes between IMRT to proton therapy.
Change in patient reported outcomes (PRO) as assessed by MDASI-BT | Baseline up to 60 months
  Will use a 2-sample t-test with a one-sided significance level of 0.05, with a Bonferroni adjustment to account for the neurocognitive function and symptom assessments resulting in an overall type I error of 0.1, there will be 72% statistical power to detect a medium effect size of 0.5 standard deviation for a comparison of the change from baseline to 6 months after randomization between the experimental and the control arm. Will compare PRO outcomes between IMRT to proton therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Vogelbaum, Principal Investigator — NRG Oncology
Locations (214):
- United States (197):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Piedmont Newnan Hospital, Newnan, Georgia
  - Piedmont Henry Hospital, Stockbridge, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - ProCure Proton Therapy Center-Somerset, Somerset, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Westchester Medical Center, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Tata Memorial Hospital, Mumbai, India
- Japan (7):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Keio University, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia